CLINICAL TRIAL: NCT06099132
Title: Antagonist Activation Measurement at the Ankle Using High-density and Bipolar Surface EMG in Chronic Hemiparesis
Acronym: CC2017
Status: Completed | Type: Observational
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Emilie Hutin, Director, Henri Mondor University Hospital
Other Study IDs: CC2017
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Muscle Hypertonia; Spasticity, Muscle
MeSH Terms: conditions — Stroke; Muscle Hypertonia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electromyographic measurements — HD and bipolar EMG were assessed from gastrocnemius medialis (GM), soleus (SO) and tibialis anterior (TA) at seated position, ankle at 0°, during isometric submaximal effort and maximal effort, knee flexed (90°) and knee extended (0°)

SUMMARY:
In chronic hemiparesis, abnormal antagonist muscle activation in the paretic lower limb contributes to impair ambulation capacities. A biased estimate of antagonist muscle activation when using surface bipolar EMG compared with high-density (HD) EMG has been previously reported in healthy subjects. The present study compares muscles cocontraction at the paretic ankle estimated with a pair of and multi-channel surface EMG.

DETAILED DESCRIPTION:
In chronic hemiparesis, gait velocity deficit is associated with a disturbed voluntary movement caused especially by inappropriate antagonist muscle activation. The present study investigates muscles cocontraction at the paretic ankle estimated with a pair of and multi-channel surface EMG (HD-EMG) in patients after stroke. HD-EMGs were collected from gastrocnemius medialis (GM), tibialis anterior (TA) and soleus (SO) during isometric contractions. From these EMGs the study asked whether bipolar and HD-EMGs provided comparable estimates of antagonist activation. Two active contraction levels (submaximal vs. maximal) and knee positions (flexed vs. extended) were assessed for each muscle. Notwithstanding the evidence of localized antagonist activation in the GM muscle of healthy subjects, hypothesizing equally localized antagonist activation in the paretic limb may not follow from the current literature. In virtue of evidence supporting the enlargement of motor unit territories in paretic and hyperactive muscles, it may be that stroke survivors have lost their ability to regionally and appropriately activate their muscle. In this case, bipolar and HD-EMG would be expected to provide comparable antagonist activation coefficients.

ELIGIBILITY:
Inclusion Criteria:

* hemiparesis due to a non-evolutive central nervous system lesion
* time since lesion ≥ 6 months
* ability to walk 10 meters barefoot without any assistance
* cognitive abilities to understand the verbal instructions for the test according to the investigator's judgment
* absence of botulinum toxin injections within the last 3 months prior to enrolment

Exclusion Criteria:

* botulinum toxin injections within the last 3 months prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Person with chronic hemiparesis due to a non-evolutive central nervous system lesion
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Coefficient of ANtagonist activation | 5 seconds
  The Coefficient of ANtagonist activation of 3 muscles was calculated by the ratio between the root mean square amplitude during antagonist effort and maximal agonist effort for the same muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Hutin, Study Director — Hôpitaux Universitaires Henri Mondor

IPD SHARING:
Plan to Share IPD: No